CLINICAL TRIAL: NCT01749735
Title: The Effect of Transcranial Direct Current Stimulation Combined With Functional Task Training on Motor Recovery in Traumatic Brain Injury Survivors
Brief Title: Transcranial Direct Current Stimulation (tDCS) and Motor Training for Traumatic Brain Injury (TBI) Survivors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated because of lack of funding.
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Paolo Bonato, Director, Motion Analysis Lab, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009-P-000700
Record Dates: First submitted 2011-12-06; First posted 2012-12-17 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-03

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Armeo training with continuous tDCS (Experimental): Subjects will receive 10 sessions of transcranial Direct Current Stimulation (tDCS)/Armeo training over 2 weeks. Training sessions will last for 40 minutes and will focus on repetitive tasks using the Armeo device that. To deliver the stimulation, the anode will be placed over the primary motor cortex (M1) of the affected hemisphere, while the cathode will be placed over the unaffected M1 area. Direct current will be transferred by a saline-soaked pair of surface sponge electrode (35cm2). Continuous stimulation will be delivered at an intensity of 1mA while the subject undergoes the 40-minute Armeo motor training sessions.
  Interventions: Device: Transcranial Direct Current Stimulation; Device: Armeo training
- Armeo training with sham tDCS (Sham Comparator): Subjects will receive the same number of 40-minute training sessions (i.e. 10 sessions) as the subjects in the experimental group. Training will take place over a period of two weeks as per the experimental group. Also, electrodes will be positioned on the scalp as per the experimental group. However, for sham transcranial Direct Current Stimulation (tDCS), the current will be delivered for only 30 seconds. The current intensity will be gradually increased and decreased to diminish its perception.
  Interventions: Device: Sham Transcranial Direct Current Stimulation; Device: Armeo training

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Continuous mild transcranial direct current stimulation will be used while the participant plays video games using the Armeo Spring Robot to support the affected arm. Intervention: 40 minute training sessions, 5 days a week for 2 weeks.
  Other Names: Device name: Phoresor II Auto; Produced by: Iomed
  Arms: Armeo training with continuous tDCS
Device: Sham Transcranial Direct Current Stimulation — Sham transcranial direct current stimulation will be used while the participant focuses on repetitive tasks using the Armeo device that incorporate multidirectional reaching, grasp and release action of the hand of the affected arm. Intervention: 40 minute training sessions, 5 days a week for 2 weeks.
  Other Names: Device name: Phoresor II Auto; Produced by: Iomed
  Arms: Armeo training with sham tDCS
Device: Armeo training — Upper extremity training with the use of a weight support device and virtual reality.
  Other Names: Device: Armeo; Produced by: Hocoma

SUMMARY:
The aim of this study is to compare the effect of transcranial direct current stimulation and functional upper extremity task training to functional upper extremity task training alone. The functional upper extremity task training uses the Armeo Spring robotic arm to support the limb while playing functional task games on a computer.

Specific Aims:

1. To demonstrate that tDCS combined with upper extremity functional task training in a virtual environment is more effective than functional task training in a virtual environment with sham tDCS.
2. To compare cortico-excitatory changes following training with tDCS vs. sham stimulation, using paired- and single-pulse transcranial magnetic stimulation as a tool to measure cortical excitability.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, sham-controlled study comparing sham and continuous tDCS combined with repetitive upper extremity functional task training in a virtual environment. Subjects will be randomized to 1 of 2 groups: Armeo training with continuous tDCS, or sham tDCS through a randomization stratification approach. Subjects will be grouped into strata defined by the degree of weakness, and then randomized separately within each stratum according to a block randomization of 6 to receive Armeo training-continuous tDCS, or Armeo training-sham stimulation. Each subject will receive 10 training sessions over 2 weeks. Training sessions will last for 40 minutes and will focus on repetitive tasks using the Armeo device that incorporate multidirectional reaching, grasp and release action of the hand. We will use a variety of virtual tasks (computer games) in the training. Examples of the virtual tasks include 1) picking up objects from shelves placed against different walls of a room and placing them in a bin in the center foreground of the screen, 2) picking up eggs from a basket and cracking them over a frying pan, 3) picking up objects at a virtual supermarket and placing them in the shopping cart, 4) cleaning a stove top. In between training sessions, subjects will be encouraged to use the affected arm in daily activities. This will be assessed with the Motor Activity Log.

tDCS will be delivered by positioning the anode over the primary motor cortex (M1) of the affected hemisphere, while the cathode will be placed over the unaffected M1 area. The electrode localization method will be according to the International 10-20 Electrode Placement System for placement of EEG electrodes. This method has been validated with a frameless stereotactic system. Direct current will be transferred by a saline-soaked pair of surface sponge electrode (35cm2) and delivered by a battery-driven, constant current stimulator with a maximum output of 10mA. An intensity of 1mA will be used in this study (current density of 0.04 μA/cm2). Continuous stimulation will be delivered at an intensity of 1mA while the subject undergoes the 40-minute Armeo motor training sessions. For sham stimulation, the same parameters will be employed. However, the current will be applied for 30 seconds only. Current intensity will be gradually increased and decreased to diminish its perception.

Outcome measures will be performed prior to treatment initiation, at day 5, 10, and at follow-up week 1, 2 and 4 after the end of treatment. A rater blinded to the treatment will assess the effects of the intervention using the Jebsen-Taylor Hand Function Test and Box and Block Test.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* First-time moderate to severe TBI
* Arm weakness

Exclusion Criteria:

* History of seizures
* Major depression
* Agitated Behavior Scale >21
* Cognitive Impairment that interferes with understanding instructions
* Pregnancy
* Implants (e.g. metal plates, shunts, pacemaker)
* Participation in other upper extremity rehab or TBI study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: short description of the study — http://www.neuromodulationlab.org/index.php?option=com_content&view=article&id=22&Itemid=67

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Recruitment target (30) was not reached for this study. Inclusion/exclusion criteria were very restrictive hence making it difficult to recruit subjects.
Period: Overall Study
Arm/Group | Armeo Training With Continuous tDCS | Armeo Training With Sham tDCS
Started | 2 | 0
Completed | 1 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Armeo Training With Continuous tDCS | Armeo Training With Sham tDCS | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 2 |  | 2
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (8) |  | 52.5 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Jebsen-Taylor Hand Function Test Score From Baseline
Description: The Jebsen-Taylor Hand Function Test is a functional test consisting of 7 subtests. Each subtest requires that the subject performs a motor task (e.g. using one hand to pick up a small object positioned on a table in front of the subject). The test score is derived by measuring (using a stopwatch) the time in sec that the subject needs to complete the task. Individuals with no motor impairments typically need between 30 and 60 sec to complete the 7 subtests of the Jebsen-Taylor Hand Function Test.
Time Frame: Baseline, Day 5 (midpoint), Day 10 (endpoint), 1 wk post, 2 wks post, 4 wks post
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Armeo Training With Continuous tDCS | Armeo Training With Sham tDCS
Number analyzed (Participants) | 2 | 0
seconds
  Day 5 | -71.9 (67.9) |
  Day 10 | -79.0 (66.6) |
  1 week post | -20.1 (151.2) |
  2 weeks post | -17.4 (NA) — No follow up in one subject |
  4 weeks post | -26.9 (NA) — No follow up in one subject |

2. Primary Outcome: Change in Box and Block Test Score From Baseline
Description: The Box and Block Test is a functional test. Subjects are instructed to move small blocks from one box to a second box. The test measures the number of blocks that subjects can move during a period of 60 sec. The measurement unit for this task is the "number of blocks". Subjects with no motor impairments would typically move about 60 to 80 blocks in a period of 60 sec.
Time Frame: Baseline, Day 5 (midpoint), Day 10 (endpoint), 1 wk post, 2 wks post, 4 wks post
Measure: Mean (Standard Deviation); unit: number of blocks
Arm/Group | Armeo Training With Continuous tDCS | Armeo Training With Sham tDCS
Number analyzed (Participants) | 2 | 0
number of blocks
  Day 5 | 2.5 (3.5) |
  Day 10 | 3.5 (3.5) |
  1 week post | 3 (4.2) |
  2 weeks post | 1 (0) |
  4 weeks post | 6 (0) |

ADVERSE EVENTS:
Time Frame: No adverse events were observed
Arm/Group | Armeo Training With Continuous tDCS | Armeo Training With Sham tDCS
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 1/2 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Armeo Training With Continuous tDCS (N=2) | Armeo Training With Sham tDCS (N=0)
Arm Pain (General disorders) | 1 | 0 — One subject experienced arm pain, an expected adverse event related to the performance of rehabilitation exercises. The subject chose not to complete the final evaluation visit. The subject's physician prescribed Advil and the problem was resolved.

LIMITATIONS AND CAVEATS:
Patient 1 did not finish study (stopped in follow up week 2). Patient 2 missed 2 training sessions. Both patients received the intervention (tDCS group) according to the confidential patient log. There was no control group available for comparison.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No